CLINICAL TRIAL: NCT02668614
Title: Early Detection of Skin Cancer Using Millimetre-Wave Waveguide Reflectometers
Brief Title: Early Detection of Skin Cancer With Sensor Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSREB 107218
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Basal Cell
Keywords: Detection
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WR-22 model microwave sensor (Experimental)
  Interventions: Device: WR-22 model microwave sensor

INTERVENTIONS:
Device: WR-22 model microwave sensor

SUMMARY:
Skin cancer represents a large problem in today's healthcare setting. The majority of cancer diagnoses are attributed to malignant skin diseases including its major types: basal cell carcinoma, squamous cell carcinoma and melanoma. Early diagnoses is critical given early detection of malignant lesions largely increases chances of successful treatment. The current gold standard of diagnosis is histopathological examination of biopsied skin. Biopsies are not only invasive and expensive, they have variable positive predictive value, meaning they may often be preformed unnecessarily. As such, the investigators have developed a skin scanner, which is less bulky and expensive than existing similar technologies, as a tool to evaluate skin lesions prior to determining the need for a biopsy. Their objective is to obtain information in order to validate this skin scanner in the context of its ability to accurately identify basal cell carcinoma skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring skin biopsy for suspected basal cell carcinoma skin lesion
* 18 years of age or older

Exclusion Criteria:

-Poor english fluency, Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Positive predictive value | Immediately pre-biopsy

IPD SHARING:
Plan to Share IPD: Undecided